CLINICAL TRIAL: NCT06938191
Title: Comparison of Aquaporin -4, -5, -9 and IL-8 Levels in Gingival Crevicular Fluid, Dentin Fluid and Pulp Samples of Healthy and Acute Irreversible Pulpitis Teeth
Brief Title: Comparison of Aquaporin -4, -5, -9 and IL-8 Levels in GCF, Dentin Fluid and Pulp Samples
Status: Not yet recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ali Erdemir, Professor doctor, Kırıkkale University
Other Study IDs: 2025/05-2025.03.02
Record Dates: First submitted 2025-04-11; First posted 2025-04-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Pulpitis; Pulpitis - Irreversible; Pulp Inflammation; Healthy Pulp; Biomarkers
Keywords: healthy pulp; pulpitis; irreversible pulpitis; aquaporin-4; IL-8; aquaporin-5; aquaporin-9
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pulp group: Minimum 35 participants Procedure: Collection of GCF samples using periopaper. Collection of dentinal fluid using cellulose membrane. Collection of pulp tissue samples using a tirnerf.
- irreversible pulp group: Minimum 35 participants Procedure: Collection of GCF samples using periopaper. Collection of dentinal fluid using cellulose membrane. Collection of pulp tissue samples using a tirnerf.

SUMMARY:
This study aimed to compare the changes in AQP -4, -5, -9, and IL-8 levels in pulp tissue, GCF, and dentin fluid samples routinely obtained during the treatment of healthy and symptomatic teeth diagnosed with irreversible pulpitis and investigate whether there is a correlation between them.

A total of 70 patients aged 18-64 years with healthy (Group 1) and symptomatic irreversible pulpitis (Group 2) diagnosed at Kırıkkale University, Faculty of Dentistry, Department of Endodontics who will undergo routine root canal treatment will be included in the study, with a minimum of 35 participants for each group. Before starting treatment, DOS samples will be taken from healthy, symptomatic, irreversible pulpitis-diagnosed teeth and teeth contralateral to these teeth. A dentin fluid sample will be taken by holding the membrane on the dentin surface, and the pulp tissue will be removed and transferred to Eppendorf tubes. The treatment process will be completed by applying routine root canal procedures to the teeth. The samples' Aquaporin -4, -5, -9, and IL-8 levels will be analyzed by specific enzyme-linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
A total of 70 healthy (Group 1) and symptomatic irreversible pulpitis (Group 2) patients aged 18-64 years, who will undergo routine root canal treatment at Kırıkkale University, Faculty of Dentistry, Department of Endodontics, will be included in the study, with a minimum of 35 participants for each group. Before starting treatment, GCF samples will be taken from healthy, symptomatic, irreversible pulpitis-diagnosed teeth and teeth contralateral to these teeth. The tooth from which the GCF sample will be taken will be isolated with cotton pellets. After the supragingival plaque is carefully removed with a curette without touching the gums, the tooth will be dried with light air pressure for 10 seconds and periopaper strips will be placed in the gingival sulcus until resistance is felt. The periopaper strips will be removed from the gingival sulcus after 1 minute. While taking the samples, care should be taken not to contaminate with blood and saliva; contaminated samples will be repeated. The amount of GCF will be measured and recorded using the periotron device. The microliter equivalents of the values measured on the Periotron device will be recorded. Periopaper strips will be placed in 1.5 cc sterile eppendorf tubes. Gingival index and pocket depth measurements will be performed after GCF samples are taken to prevent irritation of periodontal tissues and blood contamination. Patients with a pocket depth of more than 4 mm will be excluded from the study.

After anesthesia with 1.8 ml articaine HCl containing 1:100000 epinephrine, the teeth will be isolated with rubber-dam disinfected with 70% alcohol. After disinfection of the tooth crowns and surrounding area with 30% hydrogen peroxide and 2.5% NaOCl, caries and existing restorations, if any, will be removed. In teeth with normal pulp, dentin fluid samples will be taken from the dentin cavity approximately 2 mm away from the pulp as calculated on radiographs. The exposed hard dentin surface will be dried with compressed air. Using a sterile press, 1 membrane per tooth will be applied to the exposed dentin for 1 minute and 1.5 mL will be transferred to a sterile eppendorf tube.

The pulp chamber ceiling will be removed with a No. 14 steel rond milling cutter using a micromotor. Using a sterile excavator and tirnerf, healthy and inflamed pulp samples will be removed and transferred to sterile eppendorf tubes to which 200 μl of Phosphate Buffer (PBS) pH:7.2 will be added.

While collecting the samples, care should be taken not to contaminate them with blood and saliva; GCF and dentin fluid samples with suspected contamination will be repeated. Patients with samples with contamination of pulp tissue or deterioration in storage conditions will be excluded from the study. GCF, dentin fluid and pulp tissue samples transferred to a 1.5 mL sterile eppendorf tube labeled with a code assigned to the patient with diagnosis and date, with low protein binding, kept immediately on ice, transferred to a freezer and kept at -20 °C. Samples will be transported from the clinic to the freezer at -80°C and stored in a freezer at -80°C to prevent denaturation until further analysis.

The treatment process will be completed by applying routine root canal procedures to the teeth. Teeth in the healthy pulp group with an indication for extraction will be extracted after the samples are taken, subjected to normal extraction procedures.

Aquaporin -4, -5, -9 and IL-8 levels of the samples will be analyzed by specific enzyme-linked immunosorbent assay (ELISA).

Data will be analyzed in computer environment with SPSS 28.0 (Statistical Package for the Social Sciences, NY, USA) statistical package program. Results will be evaluated at 95% confidence interval and p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 64 years.
* Patients without any known systemic disease.
* Patients requiring root canal treatment for prosthetic purposes (Healthy pulp group).
* Patients with third molars (wisdom teeth) indicated for extraction due to orthodontic or other clinical reasons (Healthy pulp group).
* Patients diagnosed with symptomatic irreversible pulpitis based on the criteria established by the American Association of Endodontists (AAE) (Symptomatic irreversible pulpitis group).
* Patients scheduled for routine root canal treatment at the Department of Endodontics, Faculty of Dentistry, Kırıkkale University.
* Patients who have provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients with any known systemic disease.
* Pregnant women or those suspected of being pregnant.
* Patients who have used antibiotics, anti-inflammatory drugs, or antidepressants within the past 4 weeks.
* Patients with significant dental plaque or calculus, gingival redness or bleeding, severe gingivitis, generalized periodontitis, or periodontal pockets deeper than 4 mm.
* Patients with teeth showing internal or external root resorption.
* Patients for whom complete rubber dam isolation cannot be achieved.
* Patients with teeth exhibiting signs of necrosis, apical lesions, swelling, or presence of a sinus tract.
* Patients with immature teeth presenting open apices.
* Patients with third molars (wisdom teeth) that are not fully erupted or have been previously diagnosed with pericoronitis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include patients aged 18-64 years who present to the Department of Endodontics, Faculty of Dentistry, Kırıkkale University, with an indication for root canal therapy and are diagnosed with either a healthy pulp status (Group 1) or symptomatic irreversible pulpitis (Group 2).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Aquaporin-4, Aquaporin-5 and Aquaporin-9 expression levels in pulp tissue in dentin fluid and GCF samples | Immediately after the procedure
  Levels of IL-8, AQP-4, AQP-5 and AQP-9 will be measured in dentin fluid, GCF and pulp tissue samples obtained during routine root canal treatment. The analysis will be performed using ELISA. The aim is to compare the expression levels between healthy individuals and patients with irreversible pulpitis.

SECONDARY OUTCOMES:
Correlation analysis between Aquaporin (AQP-4, AQP-5, AQP-9) and IL-8 levels in pulp tissue, dentin fluid, and GCF samples | Immediately after the procedure
  The study will assess the correlation between Aquaporin isoforms (AQP-4, AQP-5, and AQP-9) and IL-8 concentrations within and between two groups: healthy individuals and patients diagnosed with irreversible pulpitis. Correlation analyses will be conducted separately for each group, as well as comparatively across groups, using appropriate statistical methods to explore intra- and intergroup relationships among biomarkers in pulp tissue, dentin fluid, and GCF samples.

CONTACTS AND LOCATIONS:
Overall Officials: TANSU M BEŞPARMAK, PhD student, Principal Investigator — Kirikkale University, Faculty of Dentistry; ALİ ERDEMİR, PROF, Study Chair — Kirikkale University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: Undecided